CLINICAL TRIAL: NCT02558088
Title: Pharmacological Properties of Inhaled Salmeterol in Healthy Trained Males
Brief Title: Pharmacological Properties of Salmeterol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Nielsen, MSc., University of Copenhagen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WADA2013sal
Record Dates: First submitted 2015-09-12; First posted 2015-09-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Pharmacokinetics in Healthy Young Men
Keywords: salmeterol; pharmacokinetics; doping; beta2-agonists; long-acting beta2-agonists
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- salmeterol (Experimental)
  Interventions: Drug: Salmeterol

INTERVENTIONS:
Drug: Salmeterol

SUMMARY:
The objective of the study is to help establish a urinary threshold for salmeterol on the World Anti-doping Agency prohibited list, to avoid supratherapeutic of this substance in competitive sports.

Hence, there is no hypothesis as such.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-45 years
* Healthy

Exclusion Criteria:

* Chronic disease
* Smoking
* Habitual use of medicine
* Allergy towards salmeterol
* Unable to exercise on a bike ergometer

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Urine concentration of salmeterol | 0-24 hours after administration of the study drug

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, Professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Select State, Denmark